CLINICAL TRIAL: NCT00841334
Title: Adolescents Committed to Improvement of Nutrition and Physical Activity (ACTION)
Brief Title: Adolescents Committed to Nutrition and Physical Activity
Acronym: ACTION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Alberta Kong, MD, MPH, Associate Professor, University of New Mexico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 08-013; 5R21HL092533-02 (NIH)
Record Dates: First submitted 2009-02-09; First posted 2009-02-11 (Estimated); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Overweight; Obesity; Insulin Resistance
Keywords: Adolescent; Overweight; Obesity; Weight loss; Nutrition; Physical activity; Community-based participatory research; School-based; Primary Care; Motivational interviewing
MeSH Terms: conditions — Overweight; Obesity; Insulin Resistance; Weight Loss; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): ACTION
  Interventions: Behavioral: ACTION
- 2 (Active Comparator): Usual care
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: ACTION — Overweight/obese adolescents enrolled in ACTION will meet with SBHC providers over a 6 month period in one school year. SBHC providers will use Motivational Enhancement Therapy to motivate overweight/obese adolescents to adopt strategies for improving nutrition and physical activity.
  Arms: 1
Behavioral: Usual care — Overweight/obese adolescents in the second arm will receive a well child check with usual anticipatory guidance.
  Arms: 2

SUMMARY:
Community based participatory research principles will be used to create, implement and evaluate a culturally relevant and age-appropriate obesity intervention for adolescents who are overweight or obese. The intervention will be implemented through school-based health centers (SBHC) and will include clinical encounters with SBHC providers, use of Motivational Enhancement Therapy to help overweight/obese adolescents adopt healthier behaviors, and use of a community advisory council to develop obesity risk reduction strategies that will be delivered by print and digital video disc (DVD) media. To test efficacy of the ACTION intervention, overweight/obese adolescents will be recruited to either the intervention condition or the usual care condition. Students will have pre- and post- intervention measurements to assess if adolescents in the intervention condition will have improved risk factor profile for metabolic syndrome, improved nutrition and increased physical activity when compared with students in the usual care condition.

ELIGIBILITY:
Inclusion Criteria:

* greater than or equal to the 85th percentile in BMI
* in 9th through 11th grades at participating schools

Exclusion Criteria:

* BMI greater than or equal to 40
* previously diagnosed type 1 or type 2 diabetes
* blood pressure in the range of stage 2 hypertension
* medications that significantly interfere with weight

Ages: 13 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 145 (Actual)
Dates: Start 2008-05 (Actual); Primary Completion 2010-05 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
BMI percentile | 6 months

SECONDARY OUTCOMES:
Insulin resistance | 6 months
Lipids | 6 months
Dietary intake | 6 months
Blood pressure | 6 months
Physical activity | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Alberta S Kong, MD, MPH, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexio, Albuquerque, New Mexico, United States

REFERENCES:
- [Derived] Romaniuk D, Kimsa MW, Strzalka-Mrozik B, Kimsa MC, Kabiesz A, Romaniuk W, Mazurek U. Gene expression of IGF1, IGF1R, and IGFBP3 in epiretinal membranes of patients with proliferative diabetic retinopathy: preliminary study. Mediators Inflamm. 2013;2013:986217. doi: 10.1155/2013/986217. Epub 2013 Nov 28. PMID 24379526
- [Derived] Sussman AL, Montoya C, Werder O, Davis S, Wallerstein N, Kong AS. An adaptive CBPR approach to create weight management materials for a school-based health center intervention. J Obes. 2013;2013:978482. doi: 10.1155/2013/978482. Epub 2013 Jul 29. PMID 23984053
- [Derived] Kong AS, Sussman AL, Yahne C, Skipper BJ, Burge MR, Davis SM. School-based health center intervention improves body mass index in overweight and obese adolescents. J Obes. 2013;2013:575016. doi: 10.1155/2013/575016. Epub 2013 Mar 26. PMID 23589771